CLINICAL TRIAL: NCT07355647
Title: A Triple Blind Randomized Clinical Trial Comparing the Efficacy of a Desensitizing Agent Used With an In-Office Bleaching Technique
Brief Title: Efficacy of a Desensitizing Agent During In-Office Bleaching
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Patricia Pereira-Lores, Principal Investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025/01
Record Dates: First submitted 2025-12-10; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sensitivity, Tooth
Keywords: Tooth Bleaching; In-Office Bleaching; Desensitizing Agents; Tooth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — UltraEZ

STUDY DESIGN:
Intervention Model Description: Randomized, Triple-Blind, Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- UltraEZ Group (Experimental): A blinded clinician put in the patient bleaching trays the UltraEZ desensitizing gel, patients had to wear it 30 minutes before the session of in-office bleaching
  Interventions: Drug: UltraEZ
- Placebo Group (Placebo Comparator): A blinded clinician put in the patient bleaching trays the placebo desensitizing gel, patients had to wear it 30 minutes before the session of in-office bleaching
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UltraEZ — General Examination with bite-wings, dental prophylaxis, alginate impressions of both arches, creation of individualized bleaching trays and position finder trays. Application of the UltraEZ in the bleaching trays for 30 minutes. Isolation of the gingival tissues. Two applications of the bleaching agent of 20 minutes
  Arms: UltraEZ Group
Drug: Placebo — General Examination with bite-wings, dental prophylaxis, alginate impressions of both arches, creation of individualized bleaching trays and position finder trays. Application of the placebo in the bleaching trays for 30 minutes. Isolation of the gingival tissues. Two applications of the bleaching agent of 20 minutes
  Arms: Placebo Group

SUMMARY:
The main objective of this study is to evaluate if the use of a desensitizing agent (UltraEZ) during in-office bleaching treatment is effective in reducing tooth sensitivity , as well as doesn't affect the degree of tooth bleaching.

DETAILED DESCRIPTION:
1. Visit 1: Study information and delivery of informed consent. Recording of patient's medical history, general examination, and prophylaxis. Alginate impressions will be taken of the upper and lower arches for all the patients who meet the inclusion criteria. The impressions will be poured into plaster, and individualized trays will be made for each patient. A positioning guide-finder tray will be fabricated for each patient for color measurement.
2. Visit 2: Initial color measurement with a spectrophotometer and the positioning guide. Each patient will receive their individualized tray. A blinded clinical will put inside the trays the desensitizing agent (UltraEZ, Ultradent Products Inc.,South Jordan, UT,USA) or placebo. The patients had to wear it for 30 minutes. Then after a correct isolation the clinicians apply over the buccal surface from premolar to premolar of both arches the bleaching agent (Opalescence Boost 40%, Ultradent Products, South Jordan, USA).Two application of 20 minutes each. The sensitivity was recorded and patient were given a sensitivity test to record at home.
3. Visit 3: One week after the first bleaching session. Color measurement with a spectrophotometer and the positioning guide. In this visit the second bleaching session was done with the same steps as visit 2.
4. Visit 4: 15 days after the second bleaching session. Final data collection (color + patients sensitivity test)

ELIGIBILITY:
Inclusion Criteria:

* No oral os systemic pathology
* Periodontally Healthy
* No cavities
* Tooth shade of the canines A2 or darker

Exclusion Criteria:

* Adhesive restorations or protheses in the anterior region
* Enamel or dentin alterations
* Smoking habits
* Pregnant women
* Undergone prior bleaching treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Questionary of dental sensitivity | Perioperative, 1 hour postoperative, 24 hours postoperative, 48 hours postoperative
  General tooth sensitivity was assessed using a 5-point Numeric Rating Scale (NRS), where 0 = no sensitivity; 1 = mild discomfort; 2 = moderate discomfort that does not interfere with daily activities; 3 = considerable discomfort leading to avoidance of certain foods and beverages; and 4 = severe sensitivity requiring interruption of the bleaching treatment. Participants selected the numeric value that best represented their perceived level of tooth sensitivity.
  Pain intensity was recorded at the following time points:
  * Perioperative
  * 1 hour postoperatively
  * 24 hours postoperatively
  * 48 hours postoperatively

SECONDARY OUTCOMES:
Color evaluation of each patient | Baseline (Bleaching Day 1), 1 week later baseline (Before Bleaching day 2), Revision (One week after second bleaching session)
  Tooth color will be measured using a dental spectrophotometer, recording the following parameters: L (lightness, representing the shade from black to white on a scale of 0 to 100), a (color variation along the red-green axis, with positive values toward red/purple and negative values toward green/blue), b (color variation along the yellow-blue axis, with positive values toward yellow and negative values toward blue/purple), C (chroma, describing the intensity or saturation of a color, expressed on a scale from 0 to 40, where 0 indicates no saturation and 40 the maximum saturation), and hº (hue, representing the dominant wavelength of a color on a continuous circular scale from 0° to 360°).
  Color changes between visits will be calculated using the CIELab, CIEDE2000, and White Index for Dentistry (WID) formulas.
  Color measurements will be recorded at the following time points:
  * Baseline (Bleaching Day 1)
  * One week after baseline (Before Bleaching Day 2)
  * Follow-up (One week after)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine and Dentistry, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No